CLINICAL TRIAL: NCT01075139
Title: Pilot Trial of a Brief Motivational Intervention to Increase Physical Activity and Fruit/Vegetable Intake Among College Students
Brief Title: Brief Motivational Intervention to Increase Physical Activity and Fruit/Vegetable Intake
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Matthew P. Martens, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/A (unfunded trial)
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Physical Inactivity; Poor Diet
Keywords: Motivational interviewing; Physical activity; Diet
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Motivational Intervention (Experimental): Subjects in this condition met one-on-one with a counselor for 30 minutes. Subjects received personalized feedback regarding their current physical activity levels and fruit/vegetable intake. Counselors used a motivational interviewing style to try to help resolve ambivalence about changing their current behaviors.
  Interventions: Behavioral: Brief Motivational Intervention
- Educational information (Active Comparator): Subjects in this condition received general educational information about the benefits associated with physical activity and fruit/vegetable intake.
  Interventions: Behavioral: Educational information

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — 30 minute one-on-one meeting
  Arms: Brief Motivational Intervention
Behavioral: Educational information — Educational handouts/brochures
  Arms: Educational information

SUMMARY:
Research has shown that a high percentage of college students do not meet recommended national guidelines for physical activity or fruit/vegetable intake. The purpose of this study was to pilot test the short-term efficacy of a one-on-one, brief motivational intervention (BMI) designed to increase physical activity and fruit/vegetable intake. It was hypothesized that participants in the BMI condition would report greater physical activity and fruit/vegetable intake at follow-up than those in an education-only control condition.

ELIGIBILITY:
Inclusion Criteria:

* Two or fewer days of 30+ minutes of moderate physical activity per week
* Zero days of 20+ minutes of vigorous physical activity per week

Exclusion Criteria:

* Three or more days of 30+ minutes of moderate physical activity per week
* One or more days of 20+ minutes of vigorous physical activity per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Vigorous physical activity minutes per week. | One-month follow-up.

SECONDARY OUTCOMES:
Moderate physical activity minutes per week. | One-month follow-up.
Fruit and vegetable intake per week | One-month follow-up
  Number of fruit and vegetable servings per day per week

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Martens, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Memphis, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Martens MP, Buscemi J, Smith AE, Murphy JG. The short-term efficacy of a brief motivational intervention designed to increase physical activity among college students. J Phys Act Health. 2012 May;9(4):525-32. doi: 10.1123/jpah.9.4.525. Epub 2011 May 12. PMID 21934167